CLINICAL TRIAL: NCT02951351
Title: Topical Proparacaine Eye Drops to Improve the Experience of Patients Undergoing Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: VitreoRetinal Surgery, PA (Other); Research to Prevent Blindness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-004063
Record Dates: First submitted 2016-10-29; First posted 2016-11-01 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Age-related Macular Degeneration; Diabetic Macular Edema; Injection Site; Injection Site Infection; Pain, Postoperative
MeSH Terms: conditions — Macular Degeneration; Pain, Postoperative | interventions — proxymetacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard procedure + Culture (Active Comparator): Patients will undergo the standard injection protocol. A conjunctival culture will then be obtained followed by the application of povidone-iodine to the eyelashes and eyelid margins. Patients will be randomized to receive 5% povidone-iodine drop to the conjunctival surface followed by conjunctival culture then re-application of 5% povidone-iodine drop to the conjunctival surface. Injection will then proceed.
  Interventions: Procedure: Conjunctival culture
- Proparacaine + Culture (Experimental): Patients will undergo the standard injection protocol. A conjunctival culture will then be obtained followed by the application of povidone-iodine to the eyelashes and eyelid margins. Patients will undergo application of another drop of topical anesthetic followed by conjunctival culture. After the culture, this group of patients will have 5% povidone iodine applied to the conjunctival surface. Intravitreal injection will then proceed.
  Interventions: Drug: Proparacaine; Procedure: Conjunctival culture

INTERVENTIONS:
Drug: Proparacaine — Extra proparacaine will be applied to the conjunctival surface to determine its role in patient experience.
  Other Names: alcaine
  Arms: Proparacaine + Culture
Procedure: Conjunctival culture — Conjunctival cultures will be performed to ensure that the intervention does not interfere with antisepsis.

SUMMARY:
The specific aims of this study are to compare patient experience with and without a proparacaine drop after povidone iodine.

DETAILED DESCRIPTION:
To ensure the extra drop does not interfere with antisepsis, conjunctival cultures will be obtained from patients undergoing intravitreal injection before and after the application of the extra eye drop. Patients will be randomized to undergo additional topical analgesia during intravitreal injection vs. the standard amount of topical analgesia. Cultures of the eyelid/conjunctiva will be taken to ensure that the additional topical analgesia does not interfere with antisepsis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing intravitreal injection who do not have active eye infections
* greater than 18 years of age

Exclusion Criteria:

* patients younger than 18 years of age
* patients with active eye infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose S Pulido, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Isenberg SJ, Apt L, Yoshimori R, Khwarg S. Chemical preparation of the eye in ophthalmic surgery. IV. Comparison of povidone-iodine on the conjunctiva with a prophylactic antibiotic. Arch Ophthalmol. 1985 Sep;103(9):1340-2. doi: 10.1001/archopht.1985.01050090092039. PMID 2994609
- [Background] Apt L, Isenberg S, Yoshimori R, Paez JH. Chemical preparation of the eye in ophthalmic surgery. III. Effect of povidone-iodine on the conjunctiva. Arch Ophthalmol. 1984 May;102(5):728-9. doi: 10.1001/archopht.1984.01040030584025. PMID 6721765
- [Background] Oguz H, Oguz E, Karadede S, Aslan G. The antibacterial effect of topical anesthetic proparacaine on conjunctival flora. Int Ophthalmol. 1999;23(2):117-20. doi: 10.1023/a:1026567912389. PMID 11196120
- [Background] van Asten F, van Middendorp H, Verkerk S, Breukink MB, Lomme RM, Hoyng CB, Evers AW, Klevering BJ. ARE INTRAVITREAL INJECTIONS WITH ULTRATHIN 33-G NEEDLES LESS PAINFUL THAN THE COMMONLY USED 30-G NEEDLES? Retina. 2015 Sep;35(9):1778-85. doi: 10.1097/IAE.0000000000000550. PMID 25901838
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Median (Full Range); unit: years] | 78.1 [52.1 to 91.5] | 73.2 [62.0 to 87.7] | 77.3 [52.1 to 91.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
Injection drug administered [Count of Participants; unit: Participants]
  Bevacizumab | 16 | 10 | 26
  Aflibercept | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With Positive Conjunctival Culture
Description: Conjunctival samples were collected after participants received either an additional drop of proparacaine or povidone iodine. Bacterial cultures were performed from conjunctival samples by the Mayo Clinic Microbiology laboratory. Bacterial species identification was performed on any and all bacteria that grew.
Time Frame: pre-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
Participants | 1 | 1
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Non-Inferiority — By non-inferiority analysis, proparacaine was inferior to povidone iodine with a 5% margin for non-inferiority. To detect non-inferiority with one positive culture in the proparacaine group, 45 patients would be required in the proparacaine group with a 5% margin; p = 0.28, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain at the Time of Injection
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. The lower the score, the lesser the perceived pain, the higher the score, the higher the perceived pain.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 2 [0 to 8] | 1 [0 to 8]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Residual Pain From Intravitreal Injection
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. The lower the score, the lesser the residual pain, the higher the score, the higher the residual pain.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 1 [0 to 8] | 0 [0 to 8]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Overall Impression of Visit for Intravitreal Injection
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. The lower the score, the more positive impression of the visit, the higher the score, the less positive impression of the visit.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 0 [0 to 4] | 0 [0 to 8]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Impression of Pre-injection Preparations
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey consisted of 6 questions and was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. The lower the score, the more positive impression of the preparation process, the higher the score, the less positive impression of the preparation process..
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 0 [0 to 6] | 0 [0 to 5]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Comfort With Intravitreal Injection Standard Procedure
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. The lower the score, the more comfortable the subject was with the procedure, the higher the score, the less comfortable the subject was with the procedure.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 0 [0 to 8] | 0 [0 to 10]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Expectation Intravitreal Injection Will Have Negative Consequences on Subject Health
Description: Subjects were asked to complete a survey about their experience with intravitreal injections after the procedure was completed. The survey was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a positive response and 10 was a negative response. A lower score indicated subjects did not expect the injection would negatively affect their overall health. Higher scores indicated subjects expected the injection would negatively affect their overall health.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 0 [0 to 4] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Expectation the Injection Will Contribute to Curing/Improving Eye Condition
Description: Patients were asked to rate their expectation on the extent to which the intravitreal injections would contribute to curing or improving their eye condition. The question was scored on a 0 to 10 numeric rating scale (NRS) where 0 was a negative response (not at all) and 10 was a positive response (to a large extent). A low score indicated the subject did not expect the injection would contribute to curing or improving the eye condition while a high score indicated the subject did expect the injection will help to cure or improve the eye condition.
Time Frame: post-injection
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
Number analyzed (Participants) | 19 | 17
score on a scale | 8 [4 to 10] | 10 [0 to 10]
Statistical Analysis 1: Comparison: Standard Procedure + Culture vs Proparacaine + Culture; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Study treatment follow up was defined as one year following last administration of study treatment.
Arm/Group | Standard Procedure + Culture | Proparacaine + Culture
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT02951351/Prot_SAP_000.pdf